CLINICAL TRIAL: NCT01161550
Title: Phase 1 Study of Cladribine Based Induction Therapy (CLAG) With ATRA (All-Trans Retinoic Acid) and Midostaurin in Relapsed/Refractory AML
Brief Title: Cladribine Based Induction Therapy With All-Trans Retinoic Acid and Midostaurin in Relapsed/Refractory AML
Acronym: CLAG ATRA AML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-1181 / 201108160
Record Dates: First submitted 2010-07-09; First posted 2010-07-13 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; Cladribine; Cytarabine; Tretinoin; midostaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): GCSF 300 mcg SC Days 1-6
  Cladribine 5 mg/m2 IV Days 2-6
  Cytarabine 2 mg/m2 IV Days 2-6
  ATRA 15 mg/m2 PO QD Days 7-20
  Midostaurin 25 mg PO BID Days 7-20
  Interventions: Drug: Granulocyte colony-stimulating factor (G-CSF); Drug: Cladribine; Drug: Cytarabine; Drug: All-Trans Retinoic Acid (ATRA); Drug: Midostaurin
- Arm 2 (Experimental): GCSF 300 mcg SC Days 1-6
  Cladribine 5 mg/m2 IV Days 2-6
  Cytarabine 2 mg/m2 IV Days 2-6
  ATRA 15 mg/m2 PO QD Days 7-20
  Midostaurin 50 mg PO BID Days 7-20
  Interventions: Drug: Granulocyte colony-stimulating factor (G-CSF); Drug: Cladribine; Drug: Cytarabine; Drug: All-Trans Retinoic Acid (ATRA); Drug: Midostaurin

INTERVENTIONS:
Drug: Granulocyte colony-stimulating factor (G-CSF)
  Other Names: Filgrastim
Drug: Cladribine
  Other Names: Litak; Movectro
Drug: Cytarabine
  Other Names: Cytosar-U; Depocyt
Drug: All-Trans Retinoic Acid (ATRA)
  Other Names: Tretinoin
Drug: Midostaurin
  Other Names: PKC412

SUMMARY:
This study will evaluate the investigational drug Midostaurin in various doses given with ATRA and CLAG chemotherapy. Midostaurin is a FLT3 inhibitor that is activated or overexpressed in a significant proportion of AML patients. Research has shown that midostaurin and drugs like midostaurin may work better in combination with chemotherapy, like CLAG. CLAG is a combination of cladribine, cytarabine, and G-CSF which is approved by the FDA and used to treat AML.

DETAILED DESCRIPTION:
The main purpose of this study is to gather information about the use of a drug called midostaurin when given with ATRA and CLAG chemotherapy. Midostaurin is an investigational drug. It is a drug that inhibits FLT3 that is mutated or overexpressed in a significant proportion of AML patients. Research has shown that midostaurin and drugs like midostaurin may work better in combination with chemotherapy, like CLAG. ATRA is known to promote myeloid differentiation and has also been shown to augment cancer cell death in combination with chemotherapy. CLAG is a combination of cladribine, cytarabine, and G-CSF which is approved by the FDA and used to treat AML. This study will look at how safe this combination is, how you tolerate the treatment, and to see what dose of midostaurin is appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥18 of age. Because no dosing or adverse event data are currently available on the use of midostaurin in combination with ATRA and CLAG in patients <18 years of age, children are excluded from this study but will be eligible for future pediatric phase 2 combination trials.
* Patient must be diagnosed with refractory or relapsed AML. For the purpose of the study, refractory AML is defined as failure to achieve CR after 2 cycles of induction chemotherapy or persistent > 40% bone marrow blasts after one cycle of chemotherapy induction. Relapsed AML is defined as any evidence of disease recurrence after achieving CR. Early relapse is defined as relapse occurring earlier than 12 months and late relapse is defined as relapse occurring later than 12 months.
* Patient must have a Karnofsky Performance Status of ≥ 70% (unless poor performance status is related to the disease).
* Patient must have the following laboratory values:

  * AST and ALT ≤ 1.5 x Upper Limit of Normal (ULN),
  * Serum Bilirubin ≤ 1.5 x ULN,
  * Serum Creatinine ≤ 1.5 x ULN. Laboratory values can be outside this range if secondary to AML disease.
* Patient must able to understand and willing to sign a written informed consent document prior to registration on study.

Exclusion Criteria:

* Patient must not have newly diagnosed AML.
* Patient must not have acute promyelocytic leukemia
* Patient must not have known CNS leukemia
* Patient must not have a history of allergic reactions to compounds of similar chemical or biologic composition to midostaurin or other agents used in the study.
* Patient must not have any uncontrolled or intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, myocardial infarction within 6 months, poorly controlled hypertension, uncontrolled diabetes, chronic renal disease, or psychiatric illness/social situation that would limit compliance with study requirements.
* Patient must not have any condition, including the presence of laboratory abnormalities, which places him/her at unacceptable risk if s/he were to participate in the study or confounds the ability to interpret data from the study.
* Patient may not concurrently use other anti-cancer agents or treatments (with the exceptions of hydroxyurea, steroids, and leukopheresis).
* Female patients must not be pregnant or breastfeeding.
* Adults of reproductive potential must employ an effective method of birth control. Barrier contraceptives must be used throughout the study in both sexes. Women of childbearing potential must have a negative serum pregnancy test 48 hours prior to administration of midostaurin. Women considered not of childbearing potential include any of the following: no menses for at least 5 years; menses within 5 years but amenorrheic for at least 2 months and luteinizing hormone (LH) and follicular stimulating hormone (FSH) values within normal range (according to definition of postmenopausal for laboratory used); bilateral oophorectomy amenorrheic for at least 3 months.
* Patient must not have impaired cardiac function including any of the following:

  * Screening ECG with a QTc > 450 msec
  * Patients with congenital long QT syndrome
  * History or presence of sustained ventricular tachycardia
  * Any history of ventricular fibrillation or torsades de pointes
  * Bradycardia defined as HR < 50 bpm
  * Right bundle branch block + left anterior hemiblock (bifascicular block)
  * Patients with myocardial infarction or unstable angina < 6 months prior to starting study drug
  * CHF NY Heart Association class III or IV
  * Patients with an ejection fraction < 50% assessed by MUGA or ECHO scan within 14 days of Day 1.
* Patients must not have a known confirmed diagnosis of HIV infection or active viral hepatitis.
* Patient may not have received any investigational agent within 30 days prior to Day 1. Patient may not be receiving any other investigational agents while on this trial.
* Patients must not have had any surgical procedure, excluding central venous catheter placement or other minor procedures (e.g. skin biopsy) within 14 days of Day 1.
* Patients must not have any pulmonary infiltrate, including those suspected to be of infectious origin. In particular, patients with resolution of clinical symptoms of pulmonary infection but with residual pulmonary infiltrates on chest x-ray are not eligible until pulmonary infiltrates have completely resolved.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-11; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Tolerability of midostaurin + ATRA given with CLAG chemotherapy | 28 days following completion of therapy
Dose limiting toxicity (DLT) of midostaurin + ATRA with CLAG chemotherapy | 28 days following completion of therapy

SECONDARY OUTCOMES:
Response | 1 year
  To determine the response rate 3, morphologic leukemia-free state, morphologic complete remission rate (CRm), cytogenetic CR (CRc) rate, CR with incomplete blood counts 1 rate, and partial remission 48 rate (PR) of patients treated with midostaurin + ATRA given with CLAG chemotherapy
Survival | 1 year
  To determine the duration of response and survival including disease-free survival (DFS), event-free survival (EFS), and overall survival (OS) in these patients
Toxicity profile of midostaurin + ATRA | 28 days following completion of treatment
Pharmacokinetics of midostaurin | Cycle 1 Day 7, Cycle 1 Day 14, and Cycle 1 Day 20

CONTACTS AND LOCATIONS:
Overall Officials: Camille Abboud, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Ramsingh G, Westervelt P, McBride A, Stockerl-Goldstein K, Vij R, Fiala M, Uy G, Cashen A, Dipersio JF, Abboud CN. Phase I study of cladribine, cytarabine, granulocyte colony stimulating factor (CLAG regimen) and midostaurin and all-trans retinoic acid in relapsed/refractory AML. Int J Hematol. 2014 Mar;99(3):272-8. doi: 10.1007/s12185-014-1503-4. Epub 2014 Feb 2. PMID 24488798
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu